CLINICAL TRIAL: NCT00414089
Title: Efficacy and Safety of Treatment With a Single Dose of 90Y-ibritumomab Tiuxetan in Patients With Previously Untreated Low Tumor Burden Indolent Non-Hodgkin's Lymphoma
Brief Title: Efficacy and Safety of Treatment With a Single Dose of 90Y-ibritumomab Tiuxetan in Patients With Low Tumor Burden Untreated or Indolent NHL
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding will not be provided for the drug
Sponsor: AHS Cancer Control Alberta (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE-10-0100
Record Dates: First submitted 2006-12-19; First posted 2006-12-21 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2007-07

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — ibritumomab tiuxetan

INTERVENTIONS:
Drug: 90Y-ibritumomab tiuxetan (Zevalin)

SUMMARY:
The purpose of this study is to see how well Zevalin works in the treatment of low grade indolent B-cell lymphoma when given to patients who have not had any previous treatment for their lymphoma and who otherwise would be followed on a "watch & wait" policy.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed indolent lymphoma including:

  * follicular grade 1 or 2
  * small lymphocytic
  * marginal zone (nodal)
  * marginal zone (splenic)
  * mucosa associated lymphoid tissue (MALT)
* no evidence of transformation
* Stage III or IV disease
* No prior therapy
* involvement by less than 25% of bone marrow on assessment of trephine biopsy
* absolute lymphocyte count ≤ x 109/L
* platelets ≥ 150 x 109/L
* hemoglobin ≥ 100g/L
* absolute neutrophil count ≥ 1.5 x 109/L
* at least one bidimensionally measurable lesion at least 2cm by CT scanning

Exclusion Criteria:

* any other anticancer treatment for NHL
* prior radiation therapy
* prior myeloablative therapy (bone marrow or peripheral blood stem cell transplant)
* no other malignancy within the past 10 years except adequately treated non-melanoma skin tumors or carcinoma in situ of the cervix
* presence of central nervous system lymphoma
* patients known to be HIV positive
* patients with known seropositivity for Hepatitis C virus, Hepatitis B virus or other active infection uncontrolled by treatment
* patients with abnormal liver function: total bilirubin > 1.5X ULN or ALT > 2.5X ULN
* patients with abnormal renal function: serum creatinine > 2.5X ULN
* known hypersensitivity to murine antibodies or proteins
* immunotherapy during the preceding 6 months (including monoclonal antibodies, interleukins, interferon)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Response

SECONDARY OUTCOMES:
Progression free survival

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Belch, MD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada